CLINICAL TRIAL: NCT05555069
Title: The Impact of Menthol Flavoring on Switching in Adult Menthol Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nikki Nollen, PhD, MA (Other)
Responsible Party: Sponsor-Investigator, Nikki Nollen, PhD, MA, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00148382
Record Dates: First submitted 2022-09-15; First posted 2022-09-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Smoking Reduction
MeSH Terms: conditions — Smoking Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol Flavor Electronic Cigarette (Active Comparator): 400 adult cigarette smokers will receive 12 weeks of menthol-flavored electronic cigarettes.
  Interventions: Other: Menthol-flavored electronic cigarette
- Tobacco Flavor Electronic Cigarette (Active Comparator): 400 adult cigarette smokers will receive 12 weeks of tobacco-flavored electronic cigarettes.
  Interventions: Other: Tobacco-flavored electronic cigarette

INTERVENTIONS:
Other: Menthol-flavored electronic cigarette — Participants will receive 12 weeks of menthol -flavored electronic cigarettes to aid in switching from combustible cigarettes. Participants will be instructed on proper use of the electronic cigarettes, educated about electronic cigarettes and participate in motivation enhancement and substituting electronic cigarettes for cigarettes.
  Arms: Menthol Flavor Electronic Cigarette
Other: Tobacco-flavored electronic cigarette — Participants will receive 12 weeks of tobacco-flavored electronic cigarettes to aid in switching from combustible cigarettes. Participants will be instructed on proper use of the electronic cigarettes, educated about electronic cigarettes and participate in motivation enhancement and substituting electronic cigarettes for cigarettes.
  Arms: Tobacco Flavor Electronic Cigarette

SUMMARY:
This study will compare the efficacy of menthol-flavored versus tobacco-flavored 4th generation nicotine salt-based pod-system e-cigarettes in facilitating a switch from combustible cigarettes to e-cigarettes in adult menthol smokers.

DETAILED DESCRIPTION:
Menthol smokers (n=800), stratified by race, will be randomized 1:1 into a 12-week open label, non-inferiority trial comparing a 4th generation nicotine salt-based pod-system e-cigarette in menthol- versus tobacco-flavored e-liquid. Follow-up will continue through week 26. The primary outcome is rate of switching from combustible cigarettes to e-cigarettes at week 12.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age
* Smoke ≥ 5 cigarettes per day (CPD)
* Smoke menthol cigarettes for ≥ 6 months
* Verified smoker (CO >5ppm)
* Functioning telephone
* Interested in switching to E-cigarettes

Exclusion Criteria:

* Interested in quitting smoking
* Use of other tobacco products in past 30 days (i.e. cigarillos, cigars, hookah, smokeless tobacco, pipes)
* E-cigarette use on ≥ 4 of the past 30 days
* Uncontrolled hypertension: BP ≥ 180(systolic) or ≥ 105 (diastolic)
* Use of smoking cessation pharmacotherapy in the month prior to enrollment
* Pregnant, contemplating getting pregnant, or breastfeeding
* Plans to move from Kansas City during the treatment and follow-up phase
* Another household member enrolled in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who switch from cigarettes to electronic cigarettes at Week 12 | Week 12
  Complete switching is defined as exclusive use of e-cigarettes, confirmed with CO< 6ppm and predominant switching; defined as use of the e-cigarette with >50% reduction in CPD. This will compare the effectiveness of menthol versus tobacco e-cigarettes at facilitating switching at Week 12.

SECONDARY OUTCOMES:
Assessment of respiratory symptoms using spirometry | Week 12
  Spirometry summarizing forced expiratory flow (FEF) 25-75% and the American Thoracic Society Questionnaire will assess will assess acute respiratory symptoms experienced by cigarette and electronic cigarette smokers. This will help assess the tobacco harm reduction of electronic cigarettes.
Amount of e-liquid consumed | Week 12
  E-liquid consumed will be measured in both groups as a measure of acceptability of menthol versus tobacco e-cigarettes.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Nollen, PhD, Principal Investigator — University of Kanas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Missouri, United States